CLINICAL TRIAL: NCT01633177
Title: Diabetes Prevention in the Vitamin D and Omega-3 Trial
Brief Title: Study of Vitamin D and Omega-3 Supplementation for Preventing Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Aruna Das Pradhan, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 0308112690000; R01DK088078 (NIH)
Record Dates: First submitted 2012-06-26; First posted 2012-07-04 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
Keywords: vitamin D; omega-3 fatty acids; Type 2 diabetes; Oral glucose tolerance test (OGTT); Insulin sensitivity; Beta-cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils; Eicosapentaenoic Acid; Docosahexaenoic Acids; Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D and Omega-3 (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3; Drug: Omega-3 fatty acid (fish oil)
- Vitamin D and Omega-3 placebo (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3; Drug: Fish oil placebo
- Vitamin D placebo and Omega-3 (Active Comparator)
  Interventions: Drug: Omega-3 fatty acid (fish oil); Dietary Supplement: Vitamin D3 placebo
- Vitamin D placebo and Omega-3 placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D3 placebo; Drug: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day.
  Other Names: cholecalciferol
  Arms: Vitamin D and Omega-3; Vitamin D and Omega-3 placebo
Drug: Omega-3 fatty acid (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Other Names: fish oil; eicosapentaenoic acid; docosahexaenoic acid; EPA; DHA; Omacor®
  Arms: Vitamin D and Omega-3; Vitamin D placebo and Omega-3
Dietary Supplement: Vitamin D3 placebo — Vitamin D3 placebo
  Arms: Vitamin D placebo and Omega-3; Vitamin D placebo and Omega-3 placebo
Drug: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D and Omega-3 placebo; Vitamin D placebo and Omega-3 placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is an ongoing randomized clinical trial in 25,875 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among nondiabetic participants in VITAL and will examine whether vitamin D or fish oil prevent type 2 diabetes. Findings from this proposed study conducted within the VITAL trial will clarify whether vitamin D and omega-3 fatty acid supplementation reduces risk of type 2 diabetes and thus will inform public health and clinical guidelines for diabetes prevention.

DETAILED DESCRIPTION:
Emerging evidence suggests favorable effects of both vitamin D and marine omega-3 fatty acids on glucose homeostasis. Optimal vitamin D intake is essential for insulin secretion and action, and omega-3 fatty acids may reduce diabetes risk as a result of favorable effects on insulin sensitivity, endothelial function, chronic inflammation, or other metabolic abnormalities. Although the metabolic effects of vitamin D and omega-3 fatty acids show considerable promise for the primary prevention of type 2 diabetes (T2D), there are no completed, ongoing, or planned randomized clinical trials of vitamin D or omega-3 supplements that include T2D as a primary outcome in a general population.

We thus propose to utilize an NIH-funded randomized trial (1 U01 CA138962) to test the hypothesis that vitamin D and omega-3 supplementation will reduce the risk of T2D. We will further assess whether and to what extent vitamin D or omega-3 supplementation will improve insulin sensitivity and pancreatic beta-cell function in a subsample of the trial cohort. The VITamin D and OmegA-3 TriaL (VITAL) is a randomized, double-blind, placebo-controlled trial specifically designed to evaluate the benefits and risks of vitamin D3 (2,000 IU/day) and marine omega-3 fatty acid (eicosapentaenoic acid [EPA] + docosahexaenoic acid [DHA], 1g/day) supplements in the primary prevention of cancer and cardiovascular disease (CVD). The VITAL trial will aim to enroll 20,000 men and women (aged ≥50 and ≥55 years, respectively). The planned treatment duration is 5 years after a 1.5-year recruitment period. This diabetes ancillary study aims to implement an inexpensive and efficient strategy to validate self-reported incident T2D cases in the entire trial population and to collect pre- and post-intervention measures of glucose, insulin, and hemoglobin A1c (HbA1c) in a subset of participants. Two methods of diabetes case validation are proposed. First, we plan to collect detailed information about diagnostic glucose testing and anti-diabetic medication use from medical records and/or supplementary questionnaires completed by the participant's physician. Second, to complement our diabetes ascertainment process, we will also plan to retrieve additional data on diabetes diagnoses and hypoglycemic medications by linking the participants with the Centers for Medicare and Medicaid Services (CMS) database. In addition to evaluating whether the study interventions impact the onset of clinical diabetes, we propose to collect pre- and post-intervention measures of glucose, insulin, and HbA1c in a subset of the participants to reliably assess whether vitamin D or omega-3 supplementation alters insulin and glucose homeostasis. We plan to recruit 1,000 participants without prior clinical diabetes at the Clinical and Translational Science Center (CTSC) site at Brigham and Women's Hospital. A standard 2-hour oral glucose tolerance test (OGTT) and HbA1c measurements will be performed during the CTSC visits at baseline and at 2-year post-randomization.

Primary Aims:

1. To test whether vitamin D3 and/or EPA+DHA supplementation reduces the risk of T2D among all initially non-diabetic participants in the VITAL trial.
2. To test whether vitamin D3 and/or EPA+DHA supplementation improves insulin sensitivity and beta-cell function in a subset of 1,000 non-diabetic participants receiving OGTT at baseline and 2-year post-randomization.

Secondary Aims:

1. To test whether vitamin D3 and/or EPA+DHA supplementation lowers HbA1c, fasting glucose and insulin, as well as other surrogate indices of insulin sensitivity and beta-cell function as determined by the homeostasis model assessment (HOMA-IR and HOMA-%B, respectively) in our substudy.
2. To test whether vitamin D3 and EPA+DHA supplementation exerts synergistic or additive effects on the risk of T2D among all initially non-diabetic participants in the VITAL trial.
3. To test whether vitamin D3 and EPA+DHA supplementation exerts synergistic or additive effects on insulin sensitivity and beta-cell function as assessed by OGTT in our substudy.

For the above main effect estimates, we will further explore whether the effect of vitamin D3 or EPA+DHA supplementation varies by (1) age, (2) sex, (3) baseline intakes of these nutrients, (4) baseline levels of 25(OH)D (for vitamin D3), (5) race/skin pigmentation (for vitamin D3), (6) geographic region (for vitamin D3), and (7) BMI (for vitamin D3).

ELIGIBILITY:
Participants in VITAL (NCT01169259) who have no history of diabetes mellitus at baseline are eligible to participate in this ancillary study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25875 (Actual)
Dates: Start 2010-09; Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Incident type 2 diabetes | 5 years

SECONDARY OUTCOMES:
OGTT index of insulin sensitivity | 2 years
OGTT index of beta-cell function | 2 years
HbA1c levels | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yiqing Song, MD, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Division of Preventive Medicine, Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tobias DK, Pradhan AD, Duran EK, Li C, Song Y, Buring JE, Cook NR, Mora S, Manson JE. Vitamin D supplementation vs. placebo and incident type 2 diabetes in an ancillary study of the randomized Vitamin D and Omega-3 Trial. Nat Commun. 2025 Apr 8;16(1):3332. doi: 10.1038/s41467-025-58721-6. PMID 40199888